CLINICAL TRIAL: NCT00848731
Title: Phase I Trial of Inhaled Nitric Oxide to Treat Acute Pulmonary Embolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CMC_kline_iNO1.1
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2022-04-25 (Actual); Status verified 2011-06

CONDITIONS: Pulmonary Embolism
Keywords: pulmonary hypertension; venous thromboembolism
MeSH Terms: conditions — Pulmonary Embolism; Hypertension, Pulmonary; Venous Thromboembolism | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- iNO (Experimental): gaseous NO is delivered by facemask
  Interventions: Drug: nitric oxide

INTERVENTIONS:
Drug: nitric oxide — nitric oxide gas is delivered by facemask

SUMMARY:
This study will test the hypothesis that patients with acute PE and dyspnea can safely inhale NO. The secondary hypothesis is that patients who are blinded to the inhaled NO concentration will sustain subjective improvement in their perception of dyspnea based upon their reported Borg dyspnea score, during inhalation of NO.

Specific aims

1. Test if patients with acute PE and shortness of breath of severity ≥ 5 on a 0-10 scale called the Borg score can have inhaled nitric oxide administered via nasal cannula or face mask in a titration protocol that increases concentration by 5 ppm in 5 min steps to a maximum of 25 ppm.
2. We will measure the number of patients who meet an absolute safety endpoint during titration. An absolute safety endpoint requires execution of a rapid weaning protocol (2 ppm decrease per minute to 0 ppm).

   Absolute safety endpoints: Two consecutive SBP measurements more than one min apart with both readings < 80 mm Hg;SaO 2 <80% for more than 15 seconds; Patient deterioration as defined by: Clinical decision for need of inotropic or pressor support for any reason, seizure, new altered mental status, focal neurological signs suggestive of cerebral ischemia, evidence of myocardial ischemia, protracted vomiting.
3. Test if the patient-reported Borg score decreases with administration of NO. Patients will not be told any details about the timing of the titration and will not be made aware of their iNO concentration when the Borg score is assessed.

DETAILED DESCRIPTION:
We propose to enroll a total of 25 patients with recently diagnosed pulmonary embolism. Inclusion criteria will include moderate to severe shortness of breath as rated by the patient on a standard scoring system, a systolic blood pressure of >89 mm Hg unless the patient has a known prior history of low blood pressure, and blood oxygen saturation of >80%. Exclusion criteria will include: altered mental status, inability to use a nasal cannula, a large need for supplemental oxygen, pregnancy, pneumothorax, recent use of nitrate-containing medications, recent use of thrombolytic drugs, requirement for inotropic or pressor support, or a level of methemoglobin greater than 10%.

After obtaining informed consent, subjects will have blood drawn and vital signs will be obtained. They will subsequently begin to breathe oxygen and NO supplied through a nasal cannula delivered from the iNOvent device. The patients will undergo serial measurements of their blood pressure, arterial oxygen saturation and will have their serum methemoglobin level monitored via a non-invasive probe. Titration of the amount of NO delivered will be made periodically based on the patient's vital signs. If an absolute safety endpoint is reached, NO will be rapidly weaned. Based on the patient's response to NO as determined by their vital signs, a maintenance dose of NO, not to exceed 25 ppm, will be reached. Subjects will continue to receive this concentration for up to 2 hours prior to weaning. Patients will be asked once more to rate the severity of their shortness of breath and blood will be drawn just prior to weaning. Should the patient reach a safety endpoint, the NO will be weaned at an earlier timepoint.

We will determine the percentage of patients able to complete the full protocol without reaching a safety endpoint, the percent change in methemoglobin level, the trend in patient-reported shortness of breath, percent change in SBP and oxygen saturation and the number of patients who withdraw during induction for any reason.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Diagnosis of acute PE requires symptoms of PE present <14 days with CT angiography interpreted as positive for acute PE. Initial evaluation for PE must be predicated upon the investigation of new or unexplained cardiopulmonary or chest-related clinical features consistent with PE, including shortness of breath, chest pain, respiratory distress, dizziness, unexplained tachypnea, tachycardia, syncope, cough or hemoptysis. All patients must have CT chest angiography with <2 mm collimation,(36) with or without indirect venography. Pulmonary arterial opacification will be achieved with power injection of non-ionic, low osmolar contrast in an antecubital vein with a timing run; the pitch, voltage, gantry speed and other technical details appropriate for each scanner.(37;38) Images will be interpreted as positive for intrapulmonary arterial filling defect consistent with acute PE using our published definitions(37;38) by a board-certified radiologist with specialty training in body CT or emergency medicine imaging in all cases.
2. SBP (SBP)> 89 mm Hg at the time of enrollment. We will allow enrollment for a patient with an SBP < 90 mm Hg prior to enrollment, or a patient with a SBP>80 mm Hg, if the patient has a documented or patient-identified history of low blood pressure and has no symptoms of shock, as described by Jones et al.(39)
3. SaO2% >80% at time of enrollment.
4. Patients must have a Borg score greater than 4/10.

Exclusion Criteria:

1. Altered mental status such that they are unable to provide consent.
2. Inability to use a nasal cannula or face mask (e.g., anatomic defect)
3. Supplemental oxygen requirement greater than can be administered via nasal cannula or face mask in order to maintain SaO2 >80%.
4. Pregnancy
5. Pneumothorax with decompression
6. A serum mtHb greater than 10%
7. Concurrent therapies including:

   1. Viagra® (sildenafil) use within the past 24 hours
   2. Levitra® (vardenafil) use within the past 24 hours
   3. Cialis® (tadalafil) use within the past 72 hours
   4. Use nitroprusside or nitroglycerine with in the past 4 hours
   5. Concomitant use of pressor or inotropic agents
   6. Use of fibrinolytic agent with in the past 14 days
   7. Use of nitrates within the past 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Borg score | 3 hours

SECONDARY OUTCOMES:
vital signs | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jeff A Kline, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States